CLINICAL TRIAL: NCT02955706
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial to Assess the Efficacy of Acetyl-L-carnitine in Patient With Alzheimer's Disease
Brief Title: Assessment the Efficacy of Acetyl-L-carnitine in Patient With Alzheimer's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NCT_ADC_IV
Record Dates: First submitted 2016-11-02; First posted 2016-11-04 (Estimated); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Acetylcarnitine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): Acetyl-L-carnitine (DongA ST)
  Interventions: Drug: Acetyl-L-Carnitine
- placebo (Placebo Comparator): Placebo of Acetyl-L-carnitine (DongA ST)
  Interventions: Drug: Placebo of Acetyl-L-Carnitine

INTERVENTIONS:
Drug: Acetyl-L-Carnitine — TID
  Other Names: Nicetile
  Arms: Active
Drug: Placebo of Acetyl-L-Carnitine — TID
  Other Names: Placebo of Nicetile
  Arms: placebo

SUMMARY:
clinical trial to assess the efficacy of Acetyl-L-carnitine

DETAILED DESCRIPTION:
A multicenter, randomized, double-blind, placebo-controlled clinical trial to assess the efficacy of Acetyl-L-carnitine in patient with Alzheimer's disease

ELIGIBILITY:
Inclusion Criteria:

* More than 50 Years
* probable Alzheimer disease according to DSM-IV and NINCDS-ADRDA standard
* 12≤K-MMSE(screening)≤26
* be able to perform examinations
* Patient taking donepezil(5mg or 10mg/day) more than 3 months
* be able to visit to hospital with caregiver

Exclusion Criteria:

* possible or probable or definite vascular dementia according to NINDS-AIREN standard
* CNS disease(Cerebrovascular diseases, Epilepsy etc) to cause dementia
* Illiteracy
* Patient taking galantamine, memantine, rivastigmine within three months
* Patient taking brain enhancer, thyroid hormone within 4 weeks
* Patient taking Central nervous system stimulant, Antipsychotic agent, anticholinergic agent within 2 weeks
* at screenig blood test: AST, ALT≥ 3 X upper limit of normal range or Hb≤8g/dL or platelet<100,000/mm3 or Serum creatinine ≥ 3 X upper limit of normal range
* Abnormal result of Vit.B12, Syphilis serology, TSH
* Severe Depression, Schizophrenia, Alcoholism, Drug addiction
* Parkinson's disease (need to drug therapy)
* Angina, Myocardial infarction, ischemia within six months
* Head injury with sense of loss within six months
* Patient taking other IP within three months
* Hypersensitivity to IP
* Sever Hearing problems or Visual impairment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-09-29 (Actual); Study Completion 2019-01-25 (Actual)

PRIMARY OUTCOMES:
ADAS-cog | 24week

SECONDARY OUTCOMES:
K-MMSE | 12week, 24week

CONTACTS AND LOCATIONS:
Overall Officials: Seol Hee Han, MD, Principal Investigator — Konkuk University Medical Center
Locations (1):
- Konkuk university medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No